CLINICAL TRIAL: NCT02102893
Title: A Multi-center, Registration Study for Gastroenteral-Pancreatic Neuroendocrine Tumors in Taiwan
Brief Title: Gastroenteral-Pancreatic Neuroendocrine Tumors in Taiwan
Status: Completed | Type: Observational
Sponsor: National Health Research Institutes, Taiwan (Other)
Collaborators: National Taiwan University Hospital (Other); National Cheng-Kung University Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: T1214
Record Dates: First submitted 2014-02-27; First posted 2014-04-03 (Estimated); Last update posted 2022-07-29 (Actual); Status verified 2015-09

CONDITIONS: Neuroendocrine Tumors
Keywords: enroll the 600 patients in this trial
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Furthermore, the investigators will provide the check of immunohistochemical staining for the tumor tissue of GEP-NET patients, including the functioning status (insulinoma, glucagonoma, gastrinoma, VIPoma) and the degree of differentiation, the expression of SSTR2 or SSTR5 and the check of possible primary site for unknown primary NET patients. This examination will provide more accurate diagnosis for the patients and further treatment suggestion for the patients.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Neuroendocrine tumors (NETs) are neoplasms originating from neuroendocrine cells located throughout the body. They secret various peptides and cause various symptoms (carcinoid syndrome) or not. The incidence of NETs was not well-known till recently when Yao et al. and Hausa et al. published their surveys of NETs using data from the US Surveillance, Epidemiology, and End Results (SEER) program and from the Norwegian Registry of Cancer (NRC). The incidence of NETs in Taiwan by using the Taiwan Cancer Registry (TCR) data was increased from 0.3 to 1.51 per 100,000 from 1996 to 2008. The increased incidence for NET worldwide probably was partially due to the awareness and improvement of diagnostic technology. Compared with the incidence in western countries, the incidence of NET is much lower in Taiwan. And the incidence of NETs in Asian Pacific Islanders was also lower than the whites and blacks in US. Gastroenteral-pancreatic NETs (GEP-NETs), accounting for half to two thirds of all NETs, is the most common site of NETs. As the progress in the understanding of pathophysiology for GEP-NET, there are two novel targeted agents shown to be effective for the treatment of GEP-NET. Meanwhile, response to mTOR inhibitor was better for Asian than Caucasian in the phase III study using everolimus for advanced pancreatic NETs. These information suggests that there is racial difference for either genetic or environmental risk factors and these factors result in different incidence and/or clinical outcome. Currently, there is limited data for thorough epidemiologic study in Taiwan. The aim of this study is to collect clinical information for GEP-NET, and survey the prognostic factors for GEP-NET in Taiwan. the investigators suppose that this epidemiologic study would provide a database potentially to improve the diagnosis, and treatment of GEP-NET. This study plans to include 600 GEP-NET patients. NET patients diagnosed after 2011.1.1 is included in this study.

Furthermore, the investigators will provide the check of immunohistochemical staining for the tumor tissue of GEP-NET patients, including the functioning status (insulinoma, glucagonoma, gastrinoma, VIPoma) and the degree of differentiation, the expression of SSTR2 or SSTR5 and the check of possible primary site for unknown primary NET patients. This examination will provide more accurate diagnosis for the patients and further treatment suggestion for the patients.

DETAILED DESCRIPTION:
2.0 OBJECTIVES

2.1 To establish the database for GEP-NET by register the clinical presentation, diagnosis, stages, treatment and clinical outcome of GEP-NET patients.

2.2 To analyze the risk and prognostic factors of GEP-NET patients. 2.3 To make a treatment consensus for GEP-NETs

3.0 PATIENT POPULATION There are approximately 500 patients estimated to meet the inclusion criteria from 10 hospitals in Taiwan. This recruitment estimate may vary and will be flexible since no formal sample size is required.

3.1 Inclusion Criteria: 3.1.1 histologically proven GEP-NET patients, according to the WHO classification in any stage.

3.1.2 Signed informed consent 3.2 Exclusion criteria: 3.2.1 patients of GEP-NET without histological proof

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven GEP-NET patients, according to the WHO classification in any stage.
* Signed informed consent

Exclusion Criteria:

* Patients of GEP-NET without histological proof

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 2.1 To establish the database for GEP-NET by register the clinical presentation, diagnosis, stages, treatment and clinical outcome of GEP-NET patients.
  2.2 To analyze the risk and prognostic factors of GEP-NET patients. 2.3 To make a treatment consensus for GEP-NETs
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2014-02-13; Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

PRIMARY OUTCOMES:
To establish the database for GEP-NET by register the clinical presentation, diagnosis, stages, treatment and clinical outcome of GEP-NET patients. | There are approximately 500 patients estimated to meet the inclusion criteria from 10 hospitals in Taiwan. This recruitment estimate may vary and will be flexible since no formal sample size is required.
  Survival analysis will be conducted to calculate the hazard ratio of GEP-NET outcomes (overall survival, disease-free survival, disease-specific survival, and second primary) associated with potential prognostic factors. First, univariate survival analysis will be performed using Kaplan-Meier method. Those variables that are significantly (p<0.05) associated with GEP-NET outcomes will be included in the multivariable analysis using Cox proportional hazards regression model. With accrual interval of 10 years,an average follow-up of 5 years, and a median time to outcome of 5 years, the proposed sample size of 500 cases has a statistical power of 1.0 to detect a hazard ratio of 1.5 or more.

CONTACTS AND LOCATIONS:
Overall Officials: Li-Tzong Chen, Ph.D., Study Chair — National Institute of Cancer Research
Locations (3):
- Taiwan (3):
  - Changhua Christian Hospital, Changhua
  - Chang-Gung Memorial Hospital, Taipei
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No